CLINICAL TRIAL: NCT03840304
Title: Effectiveness of Yoga@Work Program on Neck and Shoulder Pain in Information Technology (IT) Employees
Brief Title: Effect of Yoga@Work Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Yog-Kulam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMP 0198
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Musculoskeletal Pain; Neck Pain; Shoulder Pain
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain; Shoulder Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Participants in the intervention group engaged in a 8-week yoga program delivered at their place of work (IT companies). Sessions were group-based, prescribed three sessions per week during break time (30-mins).
  Interventions: Other: Yoga@work
- Wait-list Group (No Intervention): Participants in Wait-List control were not given any intervention. 8-weeks, group followed usual break time.

INTERVENTIONS:
Other: Yoga@work — Each session included warm-up practices(for the large joints, spine, and extremities), Physical postures (Asana), breathing exercises (pranayama) and supine meditation/relaxation (savasana).
  Other Names: Yoga
  Arms: Yoga Group

SUMMARY:
Employees working in IT industry are prone to develop musculoskeletal pain,specifically back, neck and shoulder pain. This study evaluates the effectiveness of work-site yoga intervention, Yoga@work on neck and shoulder pain in IT employees.

ELIGIBILITY:
Inclusion Criteria:

* IT companies employee
* Full time employment
* Neck and Shoulder Pain
* pain of at least 3 months duration
* able to comply with intervention schedule

Exclusion Criteria:

* Pregnancy
* Refuse to give informed consent
* spinal fracture
* recent cervical spine or shoulder surgery
* recent (3 months) chemotherapy/radiotherapy/ intervention

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale for pain | change from baseline to 8 weeks
  100-mm visual analog scale (VAS), horizontal line ranging from 0mm (no pain) to 100mm (worst imaginable pain).

SECONDARY OUTCOMES:
Neck disability index (NDI) | Change from baseline to 8-weeks
  The NDI is a standard instrument for measuring self-rated disability due to neck pain.10-item, 50-point index; each of the 10 items is scored from 0 - 5. Higher points represent worse pain
Shoulder pain disability index | Change from baseline to 8-weeks
  The SPADI is a 13-item patient completed instrument. Its categories include pain (5 items) and disability (8 items), overall total scores range from 0 to 130. Higher score represent worse disability

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Study Director — Yog-Kulam; Durga Prasad Sharma, Study Chair — International Labour Organization, UN; Divya Gaur, Principal Investigator — NMP Medical Research Institute, India
Locations (1):
- NMP Medical Reserach Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided